CLINICAL TRIAL: NCT02246920
Title: A Double-Blind, Randomized, Placebo-Controlled, Parallel Group, Multi-Site Study to Compare the Therapeutic Equivalence of Fluticasone Propionate Nasal Spray, 50 mcg With Flonase® Nasal Spray in the Relief of the Signs and Symptoms of Seasonal Allergic Rhinitis
Brief Title: Clinical Equivalence Study of Fluticasone Propionate Nasal Spray, 50 mcg/Actuation vs. Flonase in Allergic Rhinitis Patients
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Development Halted
Sponsor: Teva Pharmaceuticals USA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: 71336007
Record Dates: First submitted 2014-09-18; First posted 2014-09-23 (Estimated); Results first posted 2023-06-08 (Actual); Last update posted 2023-06-08 (Actual); Status verified 2023-05

CONDITIONS: Seasonal Allergic Rhinitis
Keywords: Bioequivalence; Allergic Rhinitis
MeSH Terms: conditions — Rhinitis, Allergic, Seasonal; Rhinitis, Allergic | interventions — Fluticasone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Investigational Test Product (Experimental): Fluticasone propionate Nasal Spray, 50 mcg/actuation; 200 mcg/day for 14 days
  Interventions: Drug: Fluticasone propionate
- Reference Listed Drug (Active Comparator): Flonase® (fluticasone propionate) Nasal Spray, 50 mcg/actuation; 200 mcg/day for 14 days
  Interventions: Drug: Flonase®
- Placebo (Placebo Comparator): Saline Placebo Nasal Spray; 4 total sprays/day for 14 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Fluticasone propionate — 50 mcg/actuation Nasal Spray
  Arms: Investigational Test Product
Drug: Flonase® — 50 mcg/actuation Nasal Spray
  Other Names: Fluticasone propionate (generic name)
  Arms: Reference Listed Drug
Drug: Placebo — Inactive Nasal Spray
  Arms: Placebo

SUMMARY:
This double-blind, randomized, placebo-controlled, parallel group, multi-site study has been designed to compare the safety and efficacy of a generic Fluticasone propionate Nasal Spray, 50 mcg (Teva Pharmaceuticals USA) to the FDA Reference Listed Drug, Flonase® (fluticasone propionate) 50 mcg nasal spray (GlaxoSmithKline), in the relief of the signs and symptoms of Seasonal Allergic Rhinitis. Additionally, both the test and reference formulations will be tested for superiority against a placebo nasal spray.

ELIGIBILITY:
Inclusion Criteria:

* Male or non-pregnant, non-lactating female 12 years or age or older.
* Signed informed consent form, which meets all criteria of current FDA regulations. For patients under the age of majority in the state the study is being conducted (18 years in most states) the parent or legal guardian should sign the consent form and the child will be required to sign a patient "assent" form that will be written in such a way as to be understandable to a child.
* If female and of child-bearing potential, have a negative urine pregnancy test and is prepared to abstain from sexual intercourse or use a reliable method of contraception during the study. In order for hormonal birth control to be considered a reliable method the patient must have been on their regimen for at least 28 days.
* Documented positive allergic skin test, performed within the previous 12 months, to one or more of the allergens in season at the time the study is being conducted.
* A minimum of two consecutive years of previous history of seasonal allergic rhinitis to the pollen/allergen in season at the time the study is being conducted.
* A score of at least 6 on the reflective Total Nasal Symptom Score (rTNSS) and a minimum score of at least 2 for "nasal congestion" and a minimum score of at least 2 for one of the remaining 3 symptoms representing the 12 hours prior to the screening visit.
* An average composite score of at least 6 on the reflective Total Nasal Symptom Score (rTNSS) and a minimum score of at least 2 for "nasal congestion" and a minimum score of at least 2 for one of the remaining 3 symptoms representing the last 3 days of the 7-day lead-in period before the randomization visit and the morning of the first day of the randomization visit.

Exclusion Criteria:

* Under 12 years of age.
* Females who are pregnant, lactating, or likely to become pregnant during the study.
* Negative or lack of documented skin allergen test (performed within the previous 12 months) to at least one of the allergens in season at the time of the study is being conducted. The results of all positive shin allergen tests should be reported.
* Patients who suffer from chronic signs and symptoms of perennial allergic rhinitis (PAR) should be excluded from the study unless the Investigator assesses that the patient's current signs and symptoms are a clear exacerbation of Seasonal Allergic Rhinitis (SAR) rather than chronic PAR.
* Patients who suffer only from perennial allergic rhinitis or seasonal allergic rhinitis to a different allergen that that in season at the time the study is conducted.
* Previous history of less than 2 years of seasonal allergic rhinitis to the pollen/allergen in season at the time the study is being conducted.
* A total score of less that 6 on the reflective Total Nasal Symptom Score (rTNSS) or a score of less than 2 for "nasal congestion" or a score of less than 2 for all 3 of the remaining symptoms.
* History of asthma over the previous 2 years that required chronic therapy. Occasional acute or mild exercise induced asthma will be allowable on the condition that the treatment of the attacks is restricted to beta-agonists only.
* Patients with nasal conditions, including infectious rhinitis, rhinitis medicamentosa, or atrophic rhinitis.
* Clinically significant nasal deformity (e.g. significantly deformed septum, nasal polyps, or ulcers) or any recent nasal surgery or trauma that has not completely healed.
* Sinus infection within the previous 30 days or history of re-occuring sinus infections.
* Patient has started immunotherapy (including topical or desensitization therapy) or changed their dose of immunotherapy within 30 days of the first dose, or is likely to have to start immunotherapy, or change their current dose during the study.
* Treatment for oral Candidiasis within 30 days of starting the study or a current Candidiasis infection.
* Upper respiratory tract infection within the previous 30 days.
* Patients with a history of tuberculosis.
* Patients with the presence of glaucoma, cataracts, ocular herpes simplex, conjunctivitis, or other eye infection not related to the diagnosis of SAR within 14 days of enrollment.
* The patient has had recent exposure (30 days) or was at risk of being exposed to chicken pox or measles.
* Patients with any untreated fungal, bacterial, or systemic viral infections within the previous 30 days.
* Use of any ophthalmic steroids within 14 days or nasal, inhaled, or systemic steroids within 30 days of the study start.
* Use of medications that significantly inhibit the cytochrome P450 subfamily enzyme CYP3A4.
* Use of intranasal or systemic second-generation anti-histamines within 10 days of enrollment.
* Use of intranasal cromolyn within 14 days of enrollment.
* Use of intranasal or systemic first-generation anti-histamines, leukotriene receptor antagonists or other nasal decongestants within 3 days of enrollment.
* Use of any tricyclic anti-depressant within 30 days of enrollment.
* Patients with attention-deficit disorder being treated with methylphenidate containing products that have not been on a stable dosing regimen for at least the 30 previous days and who cannot remain on the same dosing regimen throughout the study.
* Desensitization therapy to the seasonal allergen that is causing the patients allergic rhinitis within the previous 6 months.
* Previous SAR and/or PAR that has proven unresponsive to steroid therapy.
* Any known hypersensitivity to fluticasone, other steroids, or any of the components of the study nasal sprays.
* Significant history or current evidence of chronic infectious disease, system disorder, organ disorder, or other medical condition that in the Investigator's opinion would place the study patient at undue risk by participating, or could jeopardize the integrity of the study evaluations.
* Receipt of any drug as part of a research study within 30 days prior to the first dose.
* Planned travel outside of the local area for more than 2 consecutive days or 3 days in total, during the patient's participation in the study.
* Previous participation in this study.
* The patient has a history or non-compliance with medical regimens or treatment protocols in previous clinical studies.
* The patient is a member of the investigational study staff or a member of the family of the investigational study staff.
* The patient currently smokes cigarettes, cigars, and/or pipes and is a heavy smoker (for example, on average more than 10 cigarettes per day).

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1474 (Actual)
Dates: Start 2014-03-01 (Actual); Primary Completion 2014-07-14 (Actual); Study Completion 2014-07-14 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Novum Pharmaceutical Research Services, Pittsburgh, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 1474 subjects with SAR were enrolled into placebo run-in for the study.
Pre-assignment Details: Subjects were required to enter a 7 day placebo phase prior to randomization. 296 subjects were discovered to be placebo responders and were discontinued from the trial.
Period: Overall Study
Arm/Group | Investigational Test Product | Reference Listed Drug | Placebo
Started | 484 | 460 | 234
Completed | 477 | 453 | 231
Not Completed | 7 | 7 | 3
Not completed — Adverse Event | 3 | 1 | 1
Not completed — Lost to Follow-up | 2 | 1 | 0
Not completed — Protocol Violation | 2 | 5 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Safety Population Randomized.
Groups:
- Total: Total of all reporting groups
Arm/Group | Investigational Test Product | Reference Listed Drug | Placebo | Total
Number analyzed (Participants) | 484 | 460 | 234 | 1178
Age, Continuous [Mean (Full Range); unit: years] | 39.3 [12 to 80] | 39.4 [12 to 76] | 39.1 [12 to 77] | 39.3 [12 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 292 | 274 | 154 | 720
  Male | 192 | 186 | 80 | 458
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1 | 2
  Asian | 9 | 10 | 6 | 25
  Native Hawaiian or Other Pacific Islander | 2 | 1 | 1 | 4
  Black or African American | 114 | 108 | 64 | 286
  White | 357 | 339 | 160 | 856
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 2 | 2 | 5

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Average AM/PM Reflective Total Nasal Symptom Score (rTNSS) Over Days 1 to 14.
Description: Total Nasal Symptom Score (TNSS) is defined as the sum of the patient-rated nasal symptom severity scores for the following four allergy symptoms: Runny Nose, Nasal Congestion, Itchy Nose, and Sneezing. The severity score for each symptom will be based on a 4-point scale (0 = none, 1 = mild, 2 = moderate, and 3 = severe). The higher the score, the worse the symptoms of the 4 allergy categories are (runny nose, nasal congestions, itchy nose, and sneezing.
  The primary analysis for determining the therapeutic equivalence of the Test and Reference treatments will be based on each treatment's mean change from baseline for average rTNSS over the 2 week randomization treatment period.
  The Per-Protocol Population (PPP) will be used for the primary analysis of bioequivalence.
  The Modified Intent to Treat Population (mITT) will be used for Superiority Analysis.
Time Frame: 2 week treatment period: Day 0-14
Population: Per Protocol Population
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Investigational Test Product | Reference Listed Drug | Placebo
Number analyzed (Participants) | 479 | 458 | 233
score on a scale | -1.77 (0.11) | -1.57 (0.10) | -1.26 (0.15)
Statistical Analysis 1: Comparison: Investigational Test Product vs Reference Listed Drug; Test type: Equivalence — Equivalence is established if the 90% confidence interval is contained within 80.00-125.00%; T/R Ls Mean Ratio = 108.09, 90% CI 2-sided [94.09 to 124.40]

2. Secondary Outcome: Change From Baseline in Average Instantaneous Total Nasal Symptom Score (iTNSS) Over Days 1 to 14.
Description: Secondary efficacy analysis will evaluate the mean change from baseline in average iTNSS over the 2 week randomization treatment period.
  The Per-Protocol Population (PPP) will be used for the analysis of bioequivalence.
  Total Nasal Symptom Score (TNSS) is defined as the sum of the patient-rated nasal symptom severity scores for the following four allergy symptoms: Runny Nose, Nasal Congestion, Itchy Nose, and Sneezing. The severity score for each symptom will be based on a 4-point scale (0 = none, 1 = mild, 2 = moderate, and 3 = severe). The higher the score, the worse the symptoms of the 4 allergy categories are (runny nose, nasal congestions, itchy nose, and sneezing.
Time Frame: 2 week treatment period: Day 0 to Day 14
Population: Per Protocol Population
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Investigational Test Product | Reference Listed Drug | Placebo
Number analyzed (Participants) | 479 | 458 | 233
score on a scale | -1.70 (0.11) | -1.53 (0.11) | -1.15 (0.15)
Statistical Analysis 1: Comparison: Investigational Test Product vs Reference Listed Drug; Test type: Equivalence — Equivalence is demonstrated when the 90% confidence interval is contained within 80.00-125.00%; T/R LS Mean Ratio = 107.00, 90% CI 2-sided [92.42 to 124.09]

3. Other Pre Specified Outcome: Superiority to Placebo
Description: The primary analysis for determining the superiority of each active treatment over placebo will be based on each treatment's mean change from baseline for average rTNSS over the 2 week randomization treatment period.
  The modified Intent-to-Treat Population (mITT) will be used for the primary analysis of superiority.
  Total Nasal Symptom Score (TNSS) is defined as the sum of the patient-rated nasal symptom severity scores for the following four allergy symptoms: Runny Nose, Nasal Congestion, Itchy Nose, and Sneezing. The severity score for each symptom will be based on a 4-point scale (0 = none, 1 = mild, 2 = moderate, and 3 = severe). The higher the score, the worse the symptoms of the 4 allergy categories are (runny nose, nasal congestions, itchy nose, and sneezing.
Time Frame: 2 week treatment period: Day 0 to Day 14
Population: Modified Intent to Treat
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Investigational Test Product | Reference Listed Drug | Placebo
Number analyzed (Participants) | 479 | 458 | 233
score on a scale | -1.77 (0.11) | -1.57 (0.10) | -1.26 (0.15)
Statistical Analysis 1: Comparison: Investigational Test Product vs Placebo; Test type: Superiority; p = 0.0028, ANCOVA
Statistical Analysis 2: Comparison: Reference Listed Drug vs Placebo; Test type: Superiority; p = 0.0169, ANCOVA

ADVERSE EVENTS:
Time Frame: Adverse Events were collected from the time of ICF signature through the end of the study. Total duration 4-6 weeks
Description: Subjects were queried on health status and any changes at each visit.
Arm/Group | Investigational Test Product | Reference Listed Drug | Placebo
All-Cause Mortality (participants affected / at risk) | 0/484 | 0/460 | 0/234
Serious Adverse Events (participants affected / at risk) | 2/484 | 0/460 | 0/234
Other Adverse Events (participants affected / at risk) | 0/484 | 0/460 | 0/234
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Investigational Test Product (N=484) | Reference Listed Drug (N=460) | Placebo (N=234)
Concussion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Rib Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Conversion disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI may not publish the results of this generic (ANDA) trial without sponsor review and approval.